CLINICAL TRIAL: NCT06104293
Title: Determination of Grass Pollen Allergen Concentration Inducing Rhinoconjunctivitis Symptoms in Subjects Allergic to Grass Pollen in ALYATEC Allergen Exposure Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ALY-005
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Allergic Rhinitis Due to Grass Pollen
Keywords: Allergy; Rhinitis; Pollen
MeSH Terms: conditions — Hypersensitivity; Rhinitis

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, crossover, double-blind, controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The grass pollen allergen (Phl p 5) concentrations corresponding to concentrations A, B, C and D are assigned randomly by the technician and the pharmacist of the exposure chamber so that neither the investigator, the participants nor the clinical and medical staff are aware of the exposure doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Other): Concentration A - Concentration B - Concentration C - Concentration D
  Interventions: Other: Grass Pollen Allergen Exposure
- Group 2 (Other): Concentration B - Concentration C - Concentration D - Concentration A
  Interventions: Other: Grass Pollen Allergen Exposure
- Group 3 (Other): Concentration C - Concentration D - Concentration A - Concentration B
  Interventions: Other: Grass Pollen Allergen Exposure

INTERVENTIONS:
Other: Grass Pollen Allergen Exposure — After the screening visit, subjects are randomized into 3 groups presenting a sequence of allergen concentrations with randomly defined concentrations of Ph l p 5 (0, 30, 60 and 90 ng/m3).
  Each participant undergo four different 3-hour exposure sessions to grass pollen allergen corresponding to the four different allergen concentrations.

SUMMARY:
The aim of this study is to determine the optimal concentration of grass pollen allergens inducing rhinoconjunctivitis in subjects allergic to grass pollen in ALYATEC allergen exposure chamber.

Four concentrations of grass pollen allergen (Phl p 5) are tested during 3-hour exposures: 0, 30, 60 and 90 ng/m3.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects with symptoms of allergic rhinoconjunctivitis to grass pollen without associated asthma, requiring anti-allergic treatment for at least 2 consecutive pollen seasons;
* Subjects with positive skin prick tests to grass pollen extracts (Phleum pratense): papule diameter ≥ 5 mm compared to the negative control (NaCl reaction < 2 mm));
* Subjects with Phl p 5 specific recombinant Immunoglobulin E ≥ 0.70 kIU/L;
* Forced expiratory volume in 1 second (FEV1) ≥ 70% of predicted value at screening and before allergenic exposures;
* Women of childbearing age must have a negative pregnancy test at screening and before exposure visits;

Main Exclusion Criteria:

* Specific immunotherapy (SIT) to grass pollen allergens for more than one month in the 3 years preceding the screening visit;
* Ongoing specific immunotherapy to another allergen
* History of anaphylaxis following exposure to grass pollen or grass SITs;
* Asthma
* Ear, Nose & Throat or ocular surgical intervention in the 6 months preceding inclusion;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Optimal concentration of grass allergens (Phl p 5 in ng/m3) to induce a positive rhino-conjunctivitis response in subjects allergic to grass pollen during 3 hours of exposure to grass pollen allergens in the ALYATEC Environmental Exposure Chamber (EEC) | 0 to 3 hours
  The optimal concentration of grass pollen allergens Phl p 5 in ng/m3 will be determined by evaluating the Area Under the Curve (AUC) of the rhino-conjunctivitis TSS (Total Symptoms Score).
  The value of the TSS varies from 0 (no symptom) to 24 (highest symptoms)

SECONDARY OUTCOMES:
Time to obtain a rhino-conjunctivitis response during the 3 hours of exposure to grass pollen allergens in the ALYATEC EEC | 0 to 3 hours
  The exposure time will be determined by the time necessary to obtain the first uncorrected TSS (Total Symptoms Score) score ≥ 12 and corrected ≥ 10.
  The value of the TSS varies from 0 (no symptom) to 24 (highest symptoms)
Optimal concentration of grass allergens (Phl p 5 in ng/m3) to induce a positive rhinitis response in subjects allergic to grass pollen during 3 hours of exposure to grass allergens in the ALYATEC Environmental Exposure Chamber (EEC) | 0 to 3 hours
  The optimal concentration of grass pollen allergens Phl p 5 in ng/m3 will be determined by evaluating the Area Under the Curve (AUC) of the rhinitis-related questions of the TSS (nasal congestion, rhinorrhea, nasal itching, sneezing).
  The value of the rhinitis-related questions of the TSS varies from 0 (no symptom) to 12 (highest symptoms)
Frequency of bronchial response during 3 hours of exposure in the ALYATEC EEC | 0 to 3 hours
  The frequency of bronchial response will be assessed by determining the number of subjects presenting at least one drop of FEV1 ≥ 20% during the 3 hours of exposure in ALYATEC EEC.
Use of concomitant medications during and after exposures in the EEC ALYATEC | 0 to 24 hours
  The use of concomitant medications will be assessed by determining the number of subjects using at least one treatment during and up to 24 hours after the exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- ALYATEC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ALYATEC website — https://www.alyatec.com/